CLINICAL TRIAL: NCT01399450
Title: Effectiveness of Paliperidone ER(Invega®) on Depressive Symptoms of Schizophrenia Patients: A 8-week Open-label Prospective, Non-comparative Study
Brief Title: Paliperidone ER(Invega®) on Depressive Symptoms of Schizophrenia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Yong Min Ahn, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAL-KOR-9015; PAL-KOR-9015 (Other Grant/Funding Number: Johnson and Johnson company)
Record Dates: First submitted 2011-07-20; First posted 2011-07-21 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, depressive symptom, paliperidone
MeSH Terms: conditions — Schizophrenia; Depression | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- paliperidone add on (Experimental): paliperidone add on
  Interventions: Drug: paliperidone

INTERVENTIONS:
Drug: paliperidone — paliperidone augmenting on ongoing medication
  Other Names: Invega®

SUMMARY:
The purpose of this study is changing (improving), after initiating various doses of Paliperidone ER on schizophrenia patients.

DETAILED DESCRIPTION:
In this study, investigators are going to examine the effectiveness of Paliperidone ER on depressive symptoms toward schizophrenia patients who are previously unresponsive to other oral antipsychotics. In addition, the relationship between the change of depressive symptoms and adherence will be studied. Even though this study has a limitation of being designed as an open-labelled clinical study, it would be useful for clinicians because this study examines the influences toward adherence related to various factors and the changes of depressive symptoms related to switching to Paliperidone ER, which is well-proven medication.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 ~ 65
* Patient with schizophrenia according to DSM-IV criteria
* Patient have signed on the informed consent, and well understood the objective and procedure of this study.
* Patient who need initiation of new antipsychotics due to newly-development or recurrence of acute psychosis
* MADRS≥16
* Competent patient who is manage to answer the questionnaires.
* In case of female at child-bearing age, consent to use appropriate contraceptive methods(oral pill, contraceptive injection, intrauterine device, double barrier method and contraceptive patch) during entire duration of this study.

Exclusion Criteria:

* Past history of NMS.
* Allergy or hypersensitivity to Risperidone or Paliperidone ER.
* History of using clozapine within 1 month before screening.
* Initiating or dose-changing of SSRI, MAOI, TCA within 2 months(maintenance is allowed if those have been stable for at least 30days prior to study entry and would not be any dose changes during the study).
* Initiating of Lithium, Valproic acid, Carbamazepine, Topiramate, Lamotrigine or other mood stabilizer within 2months (maintenance is allowed).
* Patient who is supposed to be impossible to participate to this study due to clinical risk of suicide or aggressive behavior based on clinician's opinion.
* History of severe gastrointestinal obstruction(pathologic or iatrogenic) or incapacity to swallow the drug form(it is not allowed to chew, divide, dissolve or make powder of clinical trial medication due to the possibility of influence on pharmacokinetics)
* Current substance dependence(DSM-IV) or past history of dependence (more than 6months)
* Significant biochemical or hematological abnormality or abnormal finding of urinalysis, based on clinician's opinion.
* History of cardiac disease which predispose to QT prolongation(sick sinus, complete AV block, CHF, ventricular tachycardia, hypokalemia or hypocalcemia) or current medication of QT prolonging drugs
* Patients who take QT prolonging drugs or have
* Pregnant or breast-feeding female patient.
* History of participating to other investigational drug trial within 1month prior to screening.
* History of taking of long-acting antipsychotics injection within 3month before screening.
* Investigator or employee at clinical trial center, personnel related to investigator or trial center on this or other study, or family of employee or investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
MADRS(montgomery asberg depression rating scale) | 8 weeks

SECONDARY OUTCOMES:
Positive and Negative Symptom Scale(PANSS) | 8 weeks
Clinical Global Impression-Schizophrenia-severity(CGI-SCH-S) | 8 weeks
Korean Drug Attitude Inventory-10 items (KDAI-10) | 8 weeks
Medication Satisfaction Questionnaire(MSQ) | 8 weeks
Clinician Rating Scale (CRS) | 8 weeks
Medication Adherence Rating Scale(MARS) | 8 weeks
Beck's Depression Inventory(BDI) | 8 weeks
Subjective Well-being Under Neuroleptic Treatment Scale(SWN) | 8 weeks
C-SSRS(Colombia-Suicide Severity Rating Scale) | 8 weeks
Clinical Laboratory Tests | 8 weeks
Liverpool University Neuroleptic Side Effect Rating Scale(LUNSERS) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yong Min Ahn, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Dongguk University International Hospital, Goyang-si
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Background] Tollefson GD, Sanger TM, Lu Y, Thieme ME. Depressive signs and symptoms in schizophrenia: a prospective blinded trial of olanzapine and haloperidol. Arch Gen Psychiatry. 1998 Mar;55(3):250-8. doi: 10.1001/archpsyc.55.3.250. PMID 9510219
- [Background] Tollefson GD, Andersen SW, Tran PV. The course of depressive symptoms in predicting relapse in schizophrenia: a double-blind, randomized comparison of olanzapine and risperidone. Biol Psychiatry. 1999 Aug 1;46(3):365-73. doi: 10.1016/s0006-3223(99)00049-9. PMID 10435202
- [Background] Emsley R, Berwaerts J, Eerdekens M, Kramer M, Lane R, Lim P, Hough D, Palumbo J. Efficacy and safety of oral paliperidone extended-release tablets in the treatment of acute schizophrenia: pooled data from three 52-week open-label studies. Int Clin Psychopharmacol. 2008 Nov;23(6):343-56. doi: 10.1097/YIC.0b013e328314e1f3. PMID 18854723
- See also: study site — http://www.snuh.org/